CLINICAL TRIAL: NCT05485740
Title: Cognitive Multisensory Rehabilitation on Upper Extremity Function in Stroke Patients
Brief Title: Cognitive Multisensory on Upper Extremity in Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Lama Saad El-Din Mahmoud, Lecturer of physical therapy, Department of Neuromuscular disorders and its surgery, faculty of physical therapy, october 6 univerisity, October 6 University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T. REC/012/003797
Record Dates: First submitted 2022-08-01; First posted 2022-08-03 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: the control group which received the selected exercise program and the study group received the same exercise training program in addition to cognitive multisensory rehabilitation program
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): the study group received the same exercise training program in addition to cognitive multisensory rehabilitation program
  Interventions: Other: cognitive multisensory rehabilitation; Other: the selected exercise program
- control group (Experimental): the control group which received the selected exercise program
  Interventions: Other: the selected exercise program

INTERVENTIONS:
Other: cognitive multisensory rehabilitation — sensorimotor rehabilitation approach, in which the patient is asked to solve sensory discrimination exercises with closed eyes or to solve multisensory discrimination exercises, e.g., by comparing feeling shapes with seeing shapes.
  Arms: study group
Other: the selected exercise program — Upper Extremity Range of motion (ROM) exercises Passive Prolonged Stretching and positioning Weight-bearing exercise

SUMMARY:
PURPOSE:

To investigate the effect of cognitive multisensory rehabilitation program on upper extremity function in stroke patients.

BACKGROUND: Cognitive Multisensory Rehabilitation (CMR) is a promising therapy for upper limb recovery in stroke, as the CMR considered an effective therapy for motor recovery for adults with stroke

DETAILED DESCRIPTION:
Thirty patients with stroke The patients will randomly be divided into two equal groups; the control group which received the selected exercise program and the study group received the same exercise training program in addition to cognitive multisensory rehabilitation program, three times per week for 2 months. The evaluation methods Action research arm test (ARAT), Fugl-Myer Assessment upper extremity (FMA-UE), manual function test and Motor Evaluation Scale for Upper Extremity

ELIGIBILITY:
Inclusion Criteria:

1. Thirty hemiplegic patients, with the onset of stroke six months or longer.
2. Both sexes, with ages ranging from 45: 60.
3. Body mass index will range from 18.5-to 29.9 Kg/m2.

Exclusion Criteria:

1. Other brain injuries/illnesses, cognitive impairment, severe sensory or proprioceptive loss.
2. Other causes of hemiplegia.
3. Other causes of upper extremity dysfunction.

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Action research arm test | 8 weeks
  one of the most commonly used upper limb outcomes that measure the activity level in stroke rehabilitation studies consists of a total of 19 functional materials and four subtests as follows: grasp, grip, pinch, and gross movement
Manual function test | 8 weeks
  is a performance-based assessment for upper limbs with paresis caused by stroke The MFT is graded on a four-level scale. The total MFT score can range from 0 (severely impaired) to 32 (full function)
Fugl Myer Assessment upper extremity | 8 weeks
  is a scale consisting of 30 items assessing motor function and 3 items assessing reflex function The FMA-UE scores of 0 through 22 represent no upper-limb capacity; scores of 23 through 31 represent poor capacity; scores of 32 through 47 represent limited capacity; scores of 48 through 52 represent notable capacity; and scores of 53 through 66 represent full upper-limb capacity, total sensation UE score 12, passive joint motion UE score 24 and UE joint pain scores 24
Motor Evaluation Scale for Upper Extremity in Stroke patients | 8 weeks
  is a scale that measures the quality of movement of the hemiparetic upper extremity The maximum total score for the MESUPES is 58. The MESUPES-arm comprises 8 items of shoulder and elbow performance, with a maximum score of 40. Each item is scored from 0 (inability to adapt muscle tone to the movement) to 5 (ability to correct and complete motion without help)

CONTACTS AND LOCATIONS:
Locations (1):
- Lama S Mahmoud, Al Jīzah, Select State, Egypt

IPD SHARING:
Plan to Share IPD: No